CLINICAL TRIAL: NCT02963623
Title: The Prediction of Postoperative Hemorrahge Amount in Total Knee Replacement Using Fibtem
Brief Title: Fibtem Predicts Postoperative Bleeding
Status: Completed | Type: Observational
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Ka Young Rhee, Associate Professor, Konkuk University Medical Center
Other Study IDs: KUH1160104
Record Dates: First submitted 2016-11-09; First posted 2016-11-15 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Postoperative Hemorrhage
Keywords: fibtem; total knee replacement
MeSH Terms: conditions — Postoperative Hemorrhage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective study to evaluate if FIBTEM predicts the amount of postoperative bleeding in total knee replacement patients.

DETAILED DESCRIPTION:
This retrospective study evaluate patients who underwent total knee replacement arthroplasty. Laboratory coagulation parameters, including FIBTEM, before anesthesia induction and after admission to the post-anesthetic care unit and decrement of postoperative haemoglobin and amount of transfusion were reviewed.

A correlation coefficient of ρ = 0.4 was calculated from a pilot study. We need at least 44 subjects with an α value of 0.05 and a power of 0.8.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent primany unilateral total knee replacement arthroplasty under general anesthesia
* patients who had FIBTEM performed

Exclusion Criteria:

* surgery under regional anaesthesia
* a simultaneous bilateral total knee replacement arthroplasty
* the second surgery of staged total knee replacement arthroplasty
* revision of total knee replacement arthroplasty
* patients who received intraoperative transfusion
* patients who use tranexamic acid
* patients who received fibrinolytic agents because of perioperative thromboembolic event
* patients who refused transfusion because of religious belief of personal causes

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: total knee replacement patients
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
haemoglobin | postoperative periods
  the decrement of haemoglobin

CONTACTS AND LOCATIONS:
Overall Officials: Ka Young LRhee, Principal Investigator — Konkuk University Medical Center
Locations (1):
- Ka Young Rhee, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes